CLINICAL TRIAL: NCT00776711
Title: An Open-Label, Randomized Phase I Study in Healthy Adults of 4 Prime-Boost Schedules With Monovalent Influenza Subunit Virion (H5N1) Vaccine (Sanofi Pasteur, Inc), Administered Alone or Following Recombinant DNA Plasmid (H5) Vaccine (VRC, NIAID)
Brief Title: Vaccine for Prevention of Bird Flu
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 090012; 09-I-0012
Record Dates: First submitted 2008-10-18; First posted 2008-10-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-01-14

CONDITIONS: Influenza, Human
Keywords: Healthy; Avian Influenza; Immunity; Preventive; Bird Flu; Healthy Volunteer; HV; Influenza
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — Vaccines

INTERVENTIONS:
Drug: Monovalent Influenza Subunit Virion (H5N1) Vaccine, A/Indonesia/05/2005
Drug: VRC-AViDNA036-00-VP

SUMMARY:
Study Design:

This is a Phase I, randomized, open-label study to evaluate the safety, tolerability, and immunogenicity of four vaccination regimens against the influenza virus hemagglutinin H5. One group will receive A/Indonesia/05/2005 (inactivated H5N1) vaccine as both prime and boost, two groups will receive the VRC-AVIDNA036-00-VP (DNA) vaccine as prime with inactivated H5N1 boost but with different boost intervals, and one group will receive the DNA vaccine twice as prime followed by H5N1 boost. The hypothesis is that these regimens will be safe for human administration and will elicit antibody and T cell responses against the H5 protein. The primary objectives are to evaluate the safety and tolerability of the investigational vaccine regimens, at a dose of 4 mg for the DNA vaccine and 90 microgram for the inactivated H5N1, in healthy adults. Secondary and exploratory objectives are related to the immunogenicity of the study vaccine regimens.

Product Description:

The inactivated H5N1 vaccine is monovalent subunit virion vaccine, A/Indonesia/05/2005 clade 2, manufactured by Sanofi Pasteur, Inc (Swiftwater, PA). Vaccine vials will be supplied at 90 microgram/0.5mL. The VRC-AVIDNA036-00-VP vaccine was developed and manufactured by VRC, NIAID and is composed of a single closed-circular DNA plasmid that encodes the H5 protein with a CMV/R promoter. Vaccine vials will be supplied at 4 mg/mL. Each vaccination will be administered intramuscularly (IM) in the deltoid muscle using needle and syringe for the H5N1 vaccine and the Biojector (Trademark) 2000 Needle-Free Injection Management System (Biojector) for the DNA vaccine.

Subjects:

A total of 60 healthy adults, ages 18-60 years will be enrolled.

Study Plan:

Subjects will be simultaneously randomized at a ratio of 1:1:1:1 into one of four groups. Subjects and clinicians will be blinded to group assignment until Day 0 following completion of the enrollment. At the point of enrollment the randomly assigned regimen will become known to subjects and clinicians. Subjects will receive either two or three injections on the schedule shown in the schema. The protocol requires five clinic visits and two telephone follow-up contacts for Groups 1, 2, and 3, and six clinic visits and three telephone follow-up contacts for Group 4.

DETAILED DESCRIPTION:
Study Design:

This is a Phase I, randomized, open-label study to evaluate the safety, tolerability, and immunogenicity of four vaccination regimens against the influenza virus hemagglutinin H5. One group will receive A/Indonesia/05/2005 (inactivated H5N1) vaccine as both prime and boost, two groups will receive the VRC-AVIDNA036-00-VP (DNA) vaccine as prime with inactivated H5N1 boost but with different boost intervals, and one group will receive the DNA vaccine twice as prime followed by H5N1 boost. The hypothesis is that these regimens will be safe for human administration and will elicit antibody and T cell responses against the H5 protein. The primary objectives are to evaluate the safety and tolerability of the investigational vaccine regimens, at a dose of 4 mg for the DNA vaccine and 90 microgram for the inactivated H5N1, in healthy adults. Secondary and exploratory objectives are related to the immunogenicity of the study vaccine regimens.

Product Description:

The inactivated H5N1 vaccine is monovalent subunit virion vaccine, A/Indonesia/05/2005 clade 2, manufactured by Sanofi Pasteur, Inc (Swiftwater, PA). Vaccine vials will be supplied at 90 microgram/0.5mL. The VRC-AVIDNA036-00-VP vaccine was developed and manufactured by VRC, NIAID and is composed of a single closed-circular DNA plasmid that encodes the H5 protein with a CMV/R promoter. Vaccine vials will be supplied at 4 mg/mL. Each vaccination will be administered intramuscularly (IM) in the deltoid muscle using needle and syringe for the H5N1 vaccine and the Biojector (Trademark) 2000 Needle-Free Injection Management System (Biojector) for the DNA vaccine.

Subjects:

A total of 60 healthy adults, ages 18-60 years will be enrolled.

Study Plan:

Subjects will be simultaneously randomized at a ratio of 1:1:1:1 into one of four groups. Subjects and clinicians will be blinded to group assignment until Day 0 following completion of the enrollment. At the point of enrollment the randomly assigned regimen will become known to subjects and clinicians. Subjects will receive either two or three injections on the schedule shown in the schema. The protocol requires five clinic visits and two telephone follow-up contacts for Groups 1, 2, and 3, and six clinic visits and three telephone follow-up contacts for Group 4.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must meet all of the following criteria:

1. 18 to 60 years old.
2. Available for clinical follow-up through Week 48.
3. If enrolling from study opening (November 2008) through June 30, 2009, immunized with the current season FDA-approved influenza vaccine prior to enrollment at the specified interval [14 days to 24 weeks prior to enrollment for the inactivated influenza vaccine OR 30 days to 24 weeks prior to enrollment for the live-attenuated influenza vaccine (FluMist (Registered Trademark))]; subjects enrolling after July 1, 2009 are not required to have prior vaccination with the most recent seasonal influenza vaccine.
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
5. Complete an AoU prior to enrollment and verbalize understanding of all questions answered incorrectly.
6. Able and willing to complete the informed consent process.
7. Willing to donate blood for sample storage to be used for future research.
8. In good general health without clinically significant medical history.
9. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than 40 within the 56 days prior to enrollment.

   Laboratory Criteria within 56 days prior to nrollment:
10. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men
11. White blood cells (WBC) = 3,300-12,000 cells/mm(3)
12. Differential either within institutional normal range or accompanied by site physician approval
13. Total lymphocyte count greater than or equal to 800 cells/mm(3)
14. Platelets = 125,000 - 500,000/mm(3)
15. Alanine aminotransferase (ALT) less than 1.25 times the upper limit of normal (ULN)
16. Serum creatinine less than or equal to 1 times the ULN (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males)
17. Negative FDA-approved HIV blood test. [Note: Results of HIV enzyme-linked immunosorbent assay (ELISA) will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study]

    Female-Specific Criteria:
18. Negative beta-HCG pregnancy test (urine or serum) for women presumed to be of reproductive potential.
19. A female subject must meet one of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

OR

Agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 28 of the study,

OR

Agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 28 of the study by one of the following methods:

* condoms, male or female, with or without a spermicide;
* diaphragm or cervical cap with spermicide;
* intrauterine device;
* contraceptive pills, patch, implant or any other FDA-approved contraceptive method;
* male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply.

Women Specific:

1. Breast-feeding or planning to become pregnant during the first 28 weeks after enrollment in the study.

   Subject has received any of the following substances:
2. Systemic immunosuppressive medications or cytotoxic medications, within the 12 weeks prior to enrollment. [With the exceptions that a short course (duration of 10 days or less or a single injection) of corticosteroids for a self-limited condition at least 2 weeks prior to enrollment in this study will not exclude study participation.]
3. Blood products within 112 days (16 weeks) prior to HIV screening
4. Immunoglobulin within 56 days (8 weeks) prior to HIV screening
5. Live attenuated vaccines within 28 days (4 weeks) prior to initial study vaccine administration
6. Investigational research agents within 28 days (4 weeks) prior to initial study vaccine administration
7. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days (2 weeks) of initial study vaccine administration
8. Current anti-TB prophylaxis or therapy
9. Previous H5 avian influenza investigational vaccine.

   Subject has a history of any of the following clinically significant conditions:
10. Contraindication to receiving an FDA approved current seasonal influenza vaccination (e.g., egg allergy)
11. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator.
12. Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
13. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
14. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
15. Thyroid disease that is not well controlled.
16. Idiopathic urticaria within the past year.
17. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
18. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
19. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
20. Seizure disorder other than: 1) febrile seizures 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
21. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
22. Allergic reaction to aminoglycoside antibiotics.
23. Guillain-Barr Syndrome.
24. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within 5 years prior to enrollment, a history of suicide plan or attempt.
25. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10-16; Primary Completion 2011-01-14 (Actual); Study Completion 2011-01-14 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AEs)

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Subbarao K, Murphy BR, Fauci AS. Development of effective vaccines against pandemic influenza. Immunity. 2006 Jan;24(1):5-9. doi: 10.1016/j.immuni.2005.12.005. PMID 16413916
- [Background] Luke CJ, Subbarao K. Vaccines for pandemic influenza. Emerg Infect Dis. 2006 Jan;12(1):66-72. doi: 10.3201/eid1201.051147. PMID 16494720
- [Background] Taubenberger JK, Reid AH, Lourens RM, Wang R, Jin G, Fanning TG. Characterization of the 1918 influenza virus polymerase genes. Nature. 2005 Oct 6;437(7060):889-93. doi: 10.1038/nature04230. PMID 16208372
- [Derived] Enama ME, Hu Z, Gordon I, Costner P, Ledgerwood JE, Grady C; VRC 306 and 307 Consent Study Teams. Randomization to standard and concise informed consent forms: development of evidence-based consent practices. Contemp Clin Trials. 2012 Sep;33(5):895-902. doi: 10.1016/j.cct.2012.04.005. Epub 2012 Apr 20. PMID 22542645
- [Derived] Ledgerwood JE, Wei CJ, Hu Z, Gordon IJ, Enama ME, Hendel CS, McTamney PM, Pearce MB, Yassine HM, Boyington JC, Bailer R, Tumpey TM, Koup RA, Mascola JR, Nabel GJ, Graham BS; VRC 306 Study Team. DNA priming and influenza vaccine immunogenicity: two phase 1 open label randomised clinical trials. Lancet Infect Dis. 2011 Dec;11(12):916-24. doi: 10.1016/S1473-3099(11)70240-7. Epub 2011 Oct 3. PMID 21975270